CLINICAL TRIAL: NCT06156124
Title: Growing up With Disabled Siblings - Opportunity or a Threat to Development? The Role of Family and Individual Factors in Going Through Adolescence - Perspective of a Healthy Child.
Brief Title: The Role of Family and Individual Factors in Going Through Adolescence - Perspective of a Healthy Child.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Gdansk (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Ariadna Łada-Maśko, Principal Investigator, University of Gdansk
Other Study IDs: 2021/41/N/HS6/00864
Record Dates: First submitted 2023-08-30; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Disability, Intellectual; Disability Psychological; Disability, Developmental; Diabetes; Sibling Relations; Adolescent Development; Adolescent Behavior; Peer Group; Well-Being, Psychological; Family Relations
Keywords: siblings; disability; teenagers; adolescence; family; adolescent crisis; development; internalizing and externalizing disorders; resiliency
MeSH Terms: conditions — Intellectual Disability; Developmental Disabilities; Diabetes Mellitus; Adolescent Behavior; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Adolescents having sibling with intellectual disability: Dyads of healthy Polish adolescents 16-18 y.o., who have sibling with intellectual disability and one of their parent. The parent's participation is necessary to assess the presence of possible disorders in a healthy child.
  Interventions: Diagnostic Test: Psychological tests and psychosocial questionnaires
- Adolescents having sibling with motor disability: Dyads of healthy Polish adolescents 16-18 y.o., who have sibling with motor disability and one of their parent. The parent's participation is necessary to assess the presence of possible disorders in a healthy child.
  Interventions: Diagnostic Test: Psychological tests and psychosocial questionnaires
- Adolescents having sibling with diabetes: Dyads of healthy Polish adolescents 16-18 y.o., who have sibling with chronic somatic disease - diabetes, and one of their parent. The parent's participation is necessary to assess the presence of possible disorders in a healthy child.
  Interventions: Diagnostic Test: Psychological tests and psychosocial questionnaires
- Adolescents having healthy sibling: Dyads of healthy Polish adolescents 16-18 y.o., who ave healthy sibling, and one of their parent. The parent's participation is necessary to assess the presence of possible disorders in a healthy child.
  Interventions: Diagnostic Test: Psychological tests and psychosocial questionnaires

INTERVENTIONS:
Diagnostic Test: Psychological tests and psychosocial questionnaires — Assessment of psychological functioning of adolescents (including occurrence of internalizing and externalizing problems, coping with adolescent crisis), family functioning (siblings relations, parental attitudes, parentification), functioning at school (school achievement, extracurricular activities), relations with peers (time spending with peers, number of friends, quality of relations). Further, the sociodemographic variables will be also measured.

SUMMARY:
The goal of this observational study is to investigate the specificity of the growing up process in young people with disabled siblings. The functioning of adolescents with disabled siblings as a person growing up in three environments will be examined: family, peers and school.

The main questions it aims to answer are:

* Does having a disabled sibling influence the functioning of a healthy child in the family system?
* Do siblings of disabled children show a higher level of maturity than their peers with properly developing siblings?
* Does having a disabled sibling modify a child's functioning among peers?
* Does having a disabled sibling modify healthy adolescent's educational experience?
* Is there a greater risk of psychological disorders among siblings of disabled children than among siblings of normally developing children?

The 160 participants' dyads will take part in the study: healthy adolescent having disabled sibling and one of his/her parents. The parents' participation is necessary to assess the presence of possible internalizing and externalizing disorders among adolescents taking part in the study. The healthy adolescent will be filling out questionnaires regarding the remaining studied variables: functioning in the family - siblings relations, parental attitudes; at school - school achievement, extracurricular activities; relations with peers - time spending with peers, number of friends, as well as the growing up process trajectory - parentification and the way of going through an adolescent crisis.

Researchers will compare four groups (40 dyads in each group): three groups of adolescents having disabled sibling 1) intellectual disability, 2) motor disability, 3) chronic somatic disease, and 4) control group - healthy adolescent having sibling without any disability, to see if they differ from each other referring to the studied variables.

DETAILED DESCRIPTION:
Background: Having a disabled sibling can be a source of extremely important and enriching experiences that foster both, the development of socio-emotional competences, as well as broaden the child's perspective and knowledge. However, the presence of the disabled child in the family, also poses many challenges for their siblings, especially in adolescence. Thus, having a disabled sibling is analysed in the literature from two main perspectives: threat and opportunity for development: 1) Children with disabled siblings often receive less attention from their parents and friends. They often experience a sense of injustice and anger, which may then result in hyperactivity, irritation and aggression manifested in school and peer functioning. Research also indicates that adolescents in this group exhibit higher levels of depression, separation anxiety, and internalizing behaviors. 2) The resource perspective, in turn, indicates a higher sense of responsibility, self-efficacy and pride in caring for sick siblings. There is less quarrel and competition among siblings, increased level of empathy, as well as an increase in self-control, tolerance and understanding are observed in siblings of children with disabilities.

Current scientific research on the functioning of families with a disabled child has focused mainly on relations with parents, parental roles, teachers, and medical staff surrounding the disabled child. The role of siblings has been limited. Therefore, the aim of the project is to investigate the specificity of the growing up process in young people with disabled siblings. The functioning of adolescents with disabled siblings as a person growing up in three environments: family, peers and school will be examined.

Participants: 160 participants' dyads will take part in the study: healthy adolescent having disabled sibling and one of his/her parents. Participants will be divided in four groups (40 dyads in each group): three groups of adolescents having disabled sibling 1) intellectual disability, 2) motor disability, 3) chronic somatic disease, and 4) control group - healthy adolescent having sibling without any disability, one of the parents will take part in the study together with every teenager.

Methodology: The proposed research model focuses both, on the difficulties associated with having a disabled sibling (e.g. possible occurrence of disorders), as well as resources (e.g. the higher quality of relationships in the family, especially in the sibling subsystem). The parents' participation is necessary to assess the presence of possible internalizing and externalizing disorders among adolescents taking part in the study. The healthy adolescent will be filling out questionnaires regarding the remaining studied variables: functioning in the family - siblings relations, parental attitudes; at school - school achievement, extracurricular activities; relations with peers - time spending with peers, number of friends, as well as the growing up process trajectory - parentification and the way of going through an adolescent crisis.

ELIGIBILITY:
Inclusion Criteria to the groups having disabled sibling:

* age between 16 and 18 years;
* having disabled sibling, depending on the group: with intellectual disability or motor disability or with chronic somatic disease (diabetes);
* participation in the study of one of the parents.

Inclusion Criteria to the group having sibling without disability (control group):

* age between 16 and 18 years;
* having healthy siblings without any disability;
* participation in the study of one of the parents.

Exclusion Criteria to the groups having disabled sibling:

* siblings with multiple disabilities, e.g. intellectual and motor disabilities.

Exclusion Criteria to the control group and groups having disabled sibling:

* being an adolescent with disability/disorder/disease;
* age below 16 and above 18 years.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Polish adolescents having sibling.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-01-12 (Estimated); Study Completion 2025-01-12 (Estimated)

PRIMARY OUTCOMES:
Siblings relations | June 13, 2023 until January 12, 2025
  Questionnaire of Relationships with Siblings. Questionnaire consist of 20 items, composed of three subscales: 1) cohesion, 2) communication, and 3) rivalry. The study participants evaluate the frequency of experiencing the given feelings and behaviors about sibling on 5-point Likert-type scale (from 1 - never, to 5 - very often).
Parental Attitudes | June 13, 2023 until January 12, 2025
  Parental Attitude Scale - 2. The questionnaire enables the evaluation of five parental attitudes: Acceptance-rejection, Demanding, Autonomy, Inconsistency, and Overprotective. The questionnaire consists of 45 items (separately for mother and father). The participants provide answers on a 5-point scale, assessing which answer best corresponds to the behavior of the mother/father towards the adolescent (from 1 - not true at all to 5 - completely true).
Relations with peers | June 13, 2023 until January 12, 2025
  Relationships with peers will be assessed on the basis of the answers given to the questions in the survey created for the purposes of the study. The questions will consider issues such as: amount of time spend with peers, number of close friends, participation in joint activities with peers. Furthermore to investigate the adolescents' quality of life in terms of relationship with peers and support from them the Polish adaptation of KidScreen-27 will be used. This questionnaire, consists of 27 items. Adolescent answers the given questions on 5-point scale (from 1 - never to 5 - always. The KidScreen-27 measures five dimensions of quality of life 1) physical well-being, 2) psychological well-being, 3) parent relationships and autonomy, 4) social support and peers, and 5) school environment. The social support and peers dimension will be used in the research.
Functioning at school | June 13, 2023 until January 12, 2025
  Functioning at school will be assessed on the basis of the answers given to the questions in the survey created for the purposes of the study. The questions will consider issues such as: school achievement (arithmetical mean grade is reported for students on the yearly certificate of class completion, in our study will be self-reported by adolescent), extracurricular activities.
Quality of life in school environment dimension | June 13, 2023 until January 12, 2025
  The Polish adaptation of KidScreen-27 will be used to investigate adolescent's quality of life in school environment dimension, which refers to adolescents' feelings towards school, their relationships with teachers and ability to concentrate and learn.
Parentification | June 13, 2023 until January 12, 2025
  Parentification Questionnaire for Youth - PQY. The self-report questionnaire captures the multidimensional nature of parentification. PQY consists of 26 items, participants rated their responses 5-point Likert-type scale (1 - never true, to 5 - always true). The scale is composed of four subscales: 1) emotional parentification toward parents, 2) instrumental parentification toward parents, 3) sense of injustice, and 4) satisfaction with the role; and additional two subscales for adolescents who have siblings: 1) instrumental parentification toward siblings, and 2) emotional parentification toward siblings. The above PQY questionnaire does not provide a total score, and score for each subscale is calculated as the mean of the ratings for the subscale items.
Adolescent crisis | June 13, 2023 until January 12, 2025
  Teenage Rebellion Questionnaire to assess one of the manifestations of the adolescent crisis - teenage rebellion. Part I describes 39 situations in which teenagers may rebel. These situations refer to three triggers (limitations, threats or discrepancies) and contain a description of a specific subject of rebellion. Part II of the questionnaire contains descriptions relating to four subject groups: 1) behaviors that are a manifestation of rebellion and the reasons for refraining from manifesting rebellion outside; 2) the judgments underlying the rebellion; 3) emotions related to rebellion; and 4) indicators on the basis of which adolescents distinguish rebellion from other mental states. The results obtained in the second part of the questionnaire make it possible to recreate the behaviors, judgments and emotions involved in adolescent rebellion that are characteristic of an individual.
Clinical problems | June 13, 2023 until January 12, 2025
  Child Behavior Checklist 6-18 (CBCL). CBCL is a widely known parent measure of emotional and behavioral problems in children and adolescents ages 6-18 years. CBCL consist of 113 items and several scales, which are arranged hierarchically. Each level of the hierarchy reflects a range of different emotional and behavioral problems. At the top of this hierarchy are the Internalizing Domain and the Externalizing Domain. The Internalizing Domain: includes three narrower scales of syndromes 1) Anxious/Depressed, 2) Withdrawn/Depressed, and 3) Somatic Complaints, whereas the Externalizing Domain includes 1) Rule Breaking Behavior and 2) Aggressive Behavior syndrome scales.

SECONDARY OUTCOMES:
Sociodemographic data | June 13, 2023 until January 12, 2025
  Authors survey of socio-demographic data including: sex, age, place of residence, school, class, parents education level and work, number of siblings (brothers and sisters separately), age of the siblings.

CONTACTS AND LOCATIONS:
Overall Officials: Ariadna B Łada-Maśko, M.A., Principal Investigator — Institute of Psychology, University of Gdansk
Locations (1):
- University of Gdansk, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided